CLINICAL TRIAL: NCT00246896
Title: A Program of Collaborative Care for Alzheimer Disease
Brief Title: Care Management for Patients With Alzheimer Disease and Their Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R01HS010884 (AHRQ)
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2005-10

CONDITIONS: Alzheimer's Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

INTERVENTIONS:
Behavioral: care management

SUMMARY:
This is a clinical trial to test the effectiveness of current guideline for the care of older adults with Alzheimer's disease. The study focuses on the primary care setting using a nurse care manager to facilitate guideline-level care. We are hypothesizing that patients who receive guideline-level care will have fewer behavioral problems than those who receive the usual care provided in primary care settings

DETAILED DESCRIPTION:
The specific aim of this proposal is to conduct a four-year randomized controlled clinical trial to test the efficacy of an integrated program of collaborative care as compared to usual care in improving the process and outcomes of care for older adults with dementia in a primary care setting. The program involves three primary components: (1) A comprehensive screening and diagnosis program in which all older adults aged 65 and older from Wishard's Community Health Centers will be screened for dementia. Patients with evidence of dementia will receive further evaluation to determine an explicit diagnosis. Roudebush VA Medical Center patients aged 65 and older with a diagnosis of dementia will receive further evaluation to determine an explicit diagnosis. (2) A multidisciplinary team approach to care for patients with dementia. This care will be coordinated through a geriatric nurse practitioner or a clinical nurse specialist working in the primary care clinic. The team includes primary care and specialist physicians, psychologist, other health care workers, and relevant social service agencies working to adhere to recommended standards of care for primary care patients with dementia. (3) A proactive longitudinal tracking program in which objective measures of process and outcomes of care are fed back to the collaborative care team so that appropriate changes in the course of therapy can be undertaken.

Although authoritative guidelines for the care of patients with Alzheimer Disease and related disorders have been published, there are no clinical trials that test the impact of close adherence to these guidelines on the outcomes of care for a group of vulnerable older adults in an urban primary care setting. We are hypothesizing that patients with dementia and their caregivers who are exposed to this program will: (1) be more likely to receive the emerging standard of care for dementia, including an explicit diagnosis of dementia and an appropriate level of evaluation, education, and management; (2) be less impaired by psychopathology and behavior disturbances; (3) be less functionally impaired at 1-year and 2-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimers Disease

Exclusion Criteria:

* Inability to understand English
* No telephone

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220
Dates: Start 2001-08; Study Completion 2005-08

PRIMARY OUTCOMES:
Neuropsychiatric Inventory
Cornell Depression in Dementia Scale
Activities of Daily Living

SECONDARY OUTCOMES:
Nursing home placement
hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M. Callahan, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Callahan CM, Boustani MA, Unverzagt FW, Austrom MG, Damush TM, Perkins AJ, Fultz BA, Hui SL, Counsell SR, Hendrie HC. Effectiveness of collaborative care for older adults with Alzheimer disease in primary care: a randomized controlled trial. JAMA. 2006 May 10;295(18):2148-57. doi: 10.1001/jama.295.18.2148. PMID 16684985